CLINICAL TRIAL: NCT00437437
Title: Phase I Study to Determine the Effect of a High Fat Meal on the Pharmacokinetics of BMS-540215, the Active Metabolite of Brivanib Alaninate in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Phase I Study to Determine the Effect of Food on Brivanib (BMS-582664)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CA182-022
Record Dates: First submitted 2007-02-14; First posted 2007-02-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Tumors
Keywords: Advanced or metastatic solid tumors
MeSH Terms: conditions — Neoplasms | interventions — brivanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Brivanib

INTERVENTIONS:
Drug: Brivanib — Tablet, Oral, Brivanib 800 mg, QD after single dose Pk comparison of food effect, until progression
  Other Names: BMS-582664

SUMMARY:
The purpose of this trial is to determine the effect of food versus a fasted state on single-dose pharmacokinetics of BMS-540215, the active metabolite of Brivanib alaninate

ELIGIBILITY:
For additional information, please contact the BMS oncology clinical trial information service at 855-216-0126 or email MyCancerStudyConnect@emergingmed.com. Please visit www.BMSStudyConnect.com for more information on clinical trial participation.

Inclusion Criteria:

* Histologic/cytologic diagnosis of advanced or metastatic solid tumors
* ECOG 0-2
* 4/6 weeks since prior therapy

Exclusion Criteria:

* Brain metastases
* Second primary malignancy
* Thromboembolic disease requiring full anticoagulation within 6 months
* Inability to swallow or absorb oral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2000-05; Primary Completion 2008-05 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To determine the effect on pharmacokinetics of BMS-540215, the active metabolite of brivanib alaninate, when administered following a high fat meal versus administration in a fasted state | throughout the study

SECONDARY OUTCOMES:
To assess safety and tolerability of Brivanib alaninate when administered in a fasted state, or following a high fat meal | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Dana-Farber Harvard Cancer Care, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Duke University Medical Center-Dept Of Medicine, Durham, North Carolina

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx